CLINICAL TRIAL: NCT06119711
Title: Micronutrient Levels and Nutritional Status in Critical Illness
Acronym: NUTRI-ICU
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Collaborators: University of Groningen (Other)
Responsible Party: Principal Investigator, Lise Beumeler, Principal Investigator, Frisius Medisch Centrum
Other Study IDs: NL83298.099.22
Record Dates: First submitted 2023-07-03; First posted 2023-11-07 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-03

CONDITIONS: Post Intensive Care Unit Syndrome; Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Short stay: Patients admitted to the ICU with a need for mechanical ventilation of less than 48 hours
  Interventions: Other: No intervention
- Long stay: Patients admitted to the ICU with a need for mechanical ventilation of 48 hours or more
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Rationale: A significant proportion of patients admitted to the Intensive Care Unit (ICU) is unable to fully recover, even when the initial cause of their illness has been treated. Inadequate dietary intake prior to admission and during the recovery phase may leave patients in a frail physical state, limiting rehabilitation potential. Commonly used methods to assess nutritional intake and nutritional status are highly impacted by various disease-related confounders and reporting bias. We hypothesise that a combined assessment of biomarkers in plasma and urine may provide a more accurate overview of nutritional status at ICU-admission.

Objective:

Main: Assess nutrition-related biomarkers in plasma and urine samples at ICU admission

Secondary:

Identify the number of micronutrient deficiencies at ICU admission Compare biomarker profile and dietary intake of short and long-stay ICU patients at baseline Compare subjective dietary intake, nutritional status and muscle thickness between patients with and without micronutrient deficiencies at baseline Study design: Observational study

Study population: Adult patients admitted to the ICU. Two groups will be recruited: patients with a short length of stay (<48 hours) and patients with a longer length of stay (≥48 hours).

Main study parameters: Biomarker status in blood and urine at ICU admission.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: In addition to standard care ICU treatment, the following measurements will be performed:

* Within 24 hours after admission blood and urine samples will be collected from existing venous line and urinary catheter
* Within 72 hours an ultrasound measurement of the upper leg will be performed.
* During ICU stay, when the patient is capable to do so, they will be asked to complete a retrospective dietary intake assessment.

The risks and negative effects of these tests are limited. However, this study asks for a time investment and physical and mental effort of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and above.

Exclusion Criteria:

* Not proficient in speaking and/or understanding Dutch
* Comorbidity highly affecting gut absorption (e.g. post-bariatric surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the ICU within six months after start of the study (March-August 2023) will be asked for consent to participate in this study. A maximum of 50 'short stay' (<48 hours admitted) patients will be included. These patients will only participate in the baseline measurements. Patients that are eligible for the standard post-ICU outpatient clinic at three months (≥48 hours admitted/ventilated) will be invited for additional study measurements at the standard care outpatient visit at three months after admission.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Number of biomarker deficits at ICU admission | at ICU admission
  Total number of biomarker deficts at ICU admission, based on data collected within 24 hours after admission on:
  Markers general health: haemoglobin (Hb), mean corpuscular volume (MCV), glucose, c-reactive protein (CRP), thyroid stimulating hormone (TSH), creatinine + glomerular filtration rate (eGFR), alanine aminotransferase (ALAT), urea, albumin, total protein, lipid profile Micronutrients: potassium, calcium, sodium, vit B11, vit B1, vit B6, vit B12, vit D, Vit C, ferritin, magnesium, chloride, phosphorus

SECONDARY OUTCOMES:
Dietary intake | at ICU admission
  24-hour dietary recall
Physical health | at ICU admission
  Bioimpedance analysis and ultrasound assessment of quadriceps muscle thickness

OTHER OUTCOMES:
Patient characteristics | at ICU admission
  Patient characteristics at ICU admission (clinical data from patient records)
Clinical data | at ICU admission
  ICU characteristics from electronic patient records

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Centre Leeuwarden, Leeuwarden, Netherlands

IPD SHARING:
Plan to Share IPD: No